CLINICAL TRIAL: NCT07161505
Title: The Efficiency of Personalized Theta-burst Stimulation for Inducing Long-lasting Changes in DLPFC
Brief Title: Personalized Theta-burst Stimulation for Long-lasting Changes in Approach/Avoidance Behavior
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: STU00223602; R00MH128454 (NIH)
Record Dates: First submitted 2025-08-26; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Approach/Avoidance Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Personalized TBS-EEG over the prefrontal cortex (Experimental): Theta burst stimulation (TBS) will be administrated with a figure-8 coil over the left dorsolateral prefrontal cortex (DLPFC) at the pulse intensity of up to 120% of the individualized resting motor threshold (rMT). Stimulation will be conducted at rest. The TBS parameters will be individualized to the prefrontal EEG activity (theta-gamma coupling) and delivered in synchrony with the prefrontal theta activity (phase). The approach/avoidance test and resting-state EEG recordings will be administered before and after the stimulation.
  Interventions: Device: TBS-EEG
- Personalized TBS-EEG over the head vertex (Active Comparator): Theta burst stimulation (TBS) will be administrated with a figure-8 coil over the postcentral gyrus (- a brain area with minimal functional relevance to the task) at the pulse intensity of up to 120% of the individualized resting motor threshold (rMT). Stimulation will be conducted at rest. The TBS parameters will be individualized to the prefrontal EEG activity (theta-gamma coupling) and delivered in synchrony with the prefrontal theta activity (phase). The approach/avoidance test and resting-state EEG recordings will be administered before and after the stimulation.
  Interventions: Device: TBS-EEG / Spatial Control
- Conventional TBS over the prefrontal cortex (Active Comparator): Theta burst stimulation (TBS) will be administrated with a figure-8 coil over the left dorsolateral prefrontal cortex (DLPFC) at the pulse intensity of up to 120% of the individualized resting motor threshold (rMT). Stimulation will be conducted at rest The TBS parameters will be randomized within the normative range of theta-gamma coupling (biomarker in the main experimental arm) and delivered in open-loop (irrespective of the EEG activity). The approach/avoidance test and resting-state EEG recordings will be administered before and after the stimulation.
  Interventions: Device: TBS / Temporal Control
- Lower intensity personalized TBS-EEG (Active Comparator): Theta burst stimulation (TBS) will be administrated with a figure-8 coil over the left dorsolateral prefrontal cortex (DLPFC) at the sub-threshold pulse intensity of up to 80% of the individualized resting motor threshold (rMT). Stimulation will be conducted at rest. The TBS parameters will be individualized to the prefrontal EEG activity (theta-gamma coupling) and delivered in synchrony with the prefrontal theta activity (phase). The approach/avoidance test and resting-state EEG recordings will be administered before and after the stimulation.
  Interventions: Device: TBS-EEG / Dose Control

INTERVENTIONS:
Device: TBS-EEG — Theta-burst stimulation (TBS) over the left dorsolateral prefrontal cortex (DLPFC) synchronized with the ongoing electroencephalographic (EEG) oscillations in the theta (3-7 Hz) range at a suprathreshold pulse intensity (up to 120% rMT).
  Arms: Personalized TBS-EEG over the prefrontal cortex
Device: TBS-EEG / Spatial Control — Theta-burst stimulation (TBS) over the postcentral gyrus, synchronized with the ongoing electroencephalographic (EEG) oscillations in the theta (3-7 Hz) range at a suprathreshold pulse intensity (up to 120% rMT).
  Arms: Personalized TBS-EEG over the head vertex
Device: TBS / Temporal Control — Theta-burst stimulation (TBS) over the left dorsolateral prefrontal cortex (DLPFC) at a suprathreshold pulse intensity (up to 120% rMT).
  Arms: Conventional TBS over the prefrontal cortex
Device: TBS-EEG / Dose Control — Theta-burst stimulation (TBS) similar to the "TBS-EEG" condition but at a subthreshold pulse intensity (up to 80% rMT).
  Arms: Lower intensity personalized TBS-EEG

SUMMARY:
This study will assess the long-lasting effects of personalized theta burst stimulation (TBS), a repetitive form of transcranial magnetic stimulation (TMS), over the left prefrontal cortex on the approach/avoidance behavior. TBS will be personalized based on the prefrontal theta rhythm captured with electroencephalography (EEG). The main questions it aims to answer are: 1. does a single session of personalized TBS synchronized with the individual theta rhythm over the left prefrontal cortex results in the outlasting changes in the individual behavior? 2. Does TBS results in the brain rhythms' changes as measured using resting-state EEG?

DETAILED DESCRIPTION:
This is a double-blinded, counterbalanced crossover study in healthy adults. Volunteers will participate in four TBS-EEG sessions. In each, the investigators will first conduct the approach/avoidance test with EEG. The TBS pulse intensity will be defined according to the resting motor threshold (rMT). After the approach/avoidance test, one of four conditions will be delivered in a randomized order: 1. Verum: personalized closed-loop TBS-EEG stimulation over the left DLPFC at a suprathreshold pulse intensity (up to 120% rMT); 2. Spatial control: personalized TBS stimulation over the functionally irrelevant postcentral gyrus, 3. Temporal control: conventional (non-personalized) TBS with random parameters but the same number of pulses over conventionally defined DLPFC. 4. Dose control: similar to verum but at a subthreshold pulse intensity (up to 80% rMT). At every session, 1,800 pulses will be applied. Following the stimulation, the participant will repeat the approach/avoidance test with EEG.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be legal adults between the ages of 18 to 65;
2. Able and willing to complete study procedures and tasks.

Exclusion Criteria:

1. History or evidence of chronic neurological or mental disorder;
2. Chronic condition that requires pharmacological treatment over the course of study participation;
3. Pregnancy or breastfeeding;
4. History or evidence of alcohol or drug addiction;
5. Contraindications for transcranial magnetic stimulation (history of seizures, metallic or electric implant in the head/neck area);
6. Contraindications for magnetic resonance imaging at 3 Tesla (non-compatible implants, metallic foreign bodies, insulin pump, pacemaker).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Approach/avoidance behavior | Within twenty minutes before and twenty minutes after the TBS procedure
  The changes in the reaction times (post-stimulation relative to pre-stimulation) for the correct responses in the approach/avoidance test.

SECONDARY OUTCOMES:
Coherence | Within twenty minutes before and twenty minutes after the TBS procedure
  The changes in the multivariate coherence in the electroencephalography (EEG) post-stimulation relative to pre-stimulation.
Theta-gamma coupling | Within twenty minutes before and twenty minutes after the TBS procedure
  The changes in the theta-gamma coupling (statistical covariation of theta and gamma oscillations) in the electroencephalography (EEG) post-stimulation relative to pre-stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Alekseichuk, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Full or partial access to trial IPD will be provided upon the request from qualified researchers at recognized research, medical, and educational institutions for educational and scientific purposes, and following execution of a data sharing agreement. The request should be sent via an institutional email and will be stored with the study materials. The request should include a short description of the scientific or educational aims.
  Fully de-identified data will be shared with the scientific community via an open repository following the publication describing the data.